CLINICAL TRIAL: NCT02906683
Title: A Phase IIa Study of TAS-303 in Female Patients With Stress Urinary Incontinence
Brief Title: Exploratory Trial of TAS-303 in Female Patients With Stress Urinary Incontinence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10060050
Record Dates: First submitted 2016-09-08; First posted 2016-09-20 (Estimated); Results first posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-05

CONDITIONS: Stress Urinary Incontinence
Keywords: Urinary Incontinence; Urinary Incontinence, Stress; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence; Lower Urinary Tract Symptoms | interventions — TAS-303

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- TAS-303 3mg (Experimental)
  Interventions: Drug: TAS-303
- TAS-303 6mg (Experimental)
  Interventions: Drug: TAS-303
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAS-303 — Oral administration for 8 weeks, once daily.
  Arms: TAS-303 3mg; TAS-303 6mg
Drug: Placebo — Oral administration for 8 weeks, once daily.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of TAS-303 in female patients with stress urinary incontinence.

DETAILED DESCRIPTION:
The main purpose of this study is to assess the efficacy of TAS-303 for 8 weeks in female patients with stress urinary incontinence (SUI) compared with placebo as measured by the percent change in incontinence episode frequency (IEF) from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Patient has symptoms of Stress Urinary Incontinence (SUI) for at least 12 weeks prior to study entry
* Patient has at least 1 incontinence episodes per day, and urinary diurnal frequency of 10 or less per day and nocturia of 2 or less per day.
* Patient is positive in 1-hour pad weight test

Exclusion Criteria:

* Patient has predominant or primary urge incontinence according to investigator judgment
* Patient had a prior surgical SUI treatment
* Patient is diagnosed stageII or more of Pelvic Organ Prolapse
* Patient has symptoms of Urinary tract infection (UTI)
* Patient is positive pregnancy test
* Patient has on physical examination, neurological and/or vaginal examination results which, in the opinion of the investigator, should exclude the subject.

Ages: 20 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taiho Pharmaceutical Co., Ltd, Study Director — Taiho Pharmaceutical Co., Ltd.
Locations (1):
- Taiho Pharmaceutical Co., Ltd selected site, Osaka, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was undertaken at 31 centers in Japan between 17 October 2016 and 25 April 2018.
  Of the 386 patients who gave informed consent and received screening tests, 49 patients were withdrawn at screening. The number of patients enrolled in the observation period was 337 patients, but after the end of the observation period, 256 patients were deemed to be eligible for enrollment in the treatment period.
Groups:
- TAS-303 3 mg: Female patients with stress urinary incontinence (SUI) orally received 3 mg of TAS-303 once daily for 8 weeks.
- TAS-303 6 mg: Female patients with SUI orally received 6 mg of TAS-303 once daily for 8 weeks.
- Placebo: Female patients with SUI orally received placebo once daily for 8 weeks.
Period: Overall Study
Arm/Group | TAS-303 3 mg | TAS-303 6 mg | Placebo
Started | 85 | 86 | 85
Completed | 84 | 81 | 82
Not Completed | 1 | 5 | 3
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 1
Not completed — Patient did not meet the eligibility criteria for the study | 1 | 0 | 0
Not completed — Study treatment becomes impossible due to changing hospital or other reasons | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Per protocol set (PPS) was used for the analysis. PPS included patients in the Full analysis set (FAS) who had no inclusion/exclusion criteria violations, received no prohibited concomitant medications or therapy; were compliant for ≥ 80% of the treatment period and completed ≥ 70% of Bladder diary at Week 8 in the treatment period. FAS included all patients who received the study drug and had ≥ 1 available efficacy endpoint before and during the treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | TAS-303 3 mg | TAS-303 6 mg | Placebo | Total
Number analyzed (Participants) | 84 | 80 | 81 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (11.8) | 56.0 (13.4) | 55.9 (11.3) | 56.3 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 80 | 81 | 245
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 84 | 80 | 81 | 245
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 84 | 80 | 81 | 245
Type of Urinary Incontinence [Count of Participants; unit: Participants]
  Stress Urinary Incontinence (SUI) | 63 | 61 | 61 | 185
  Mixed Urinary Incontinence (MUI) | 21 | 19 | 20 | 60
Prior surgery for pelvic organ prolapse [Count of Participants; unit: Participants] | 10 | 5 | 5 | 20
Urinary Incontinence episodes of <2 per 24 hours [Count of Participants; unit: Participants] | 39 | 40 | 41 | 120
Urinary Incontinence episodes of ≥2 per 24 hours [Count of Participants; unit: Participants] | 45 | 40 | 40 | 125
Number of Urinary Incontinence episodes per 24 hours [Mean (Standard Deviation); unit: episodes per 24hr] | 2.853 (2.322) | 2.499 (1.507) | 2.582 (1.673) | 2.648 (1.874)
1-hour Pad weight Test [Mean (Standard Deviation); unit: gram] — 1-hour Pad weight Test is a one hour test for measuring urinary incontinence. Patients were instructed to wear incontinence pads capable of retaining a certain amount (≥200mL) of urine leakage and to perform urinary incontinence-inducible activities (7 activities including walking and climbing stairs) for one hour. After 1-hour activity, the amount of urinary incontinence was evaluated by measuring the incontinence pad. Dryness (no incontinence) is defined as a pad weight of ≤2.0 g in this test.
  gram | 33.85 (70.98) | 29.12 (48.26) | 37.92 (60.49) | 33.65 (60.67)

OUTCOME MEASURES:

1. Primary Outcome: Incontinence Episode Frequency (IEF) Per 24 Hours at Baseline and Week 8
Time Frame: Baseline to Week 8 (8 weeks in treatment period)
Population: PPS was used for the analysis.
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | TAS-303 3 mg | TAS-303 6 mg | Placebo
Number analyzed (Participants) | 84 | 80 | 81
episodes
  IEF per 24 hours at baseline | 2.9 (2.3) | 2.5 (1.5) | 2.6 (1.7)
  IEF per 24 hours at Week 8 | 2.0 (2.3) | 1.7 (1.7) | 1.9 (1.9)

2. Primary Outcome: Mean Percentage Changes in Incontinence Episode Frequency (IEF) Per 24 Hours From Baseline to Week 8
Time Frame: Baseline to Week 8 (8 weeks in treatment period)
Population: PPS was used for the analysis.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | TAS-303 3 mg | TAS-303 6 mg | Placebo
Number analyzed (Participants) | 84 | 80 | 81
Percentage change | -34.7 (39.9) | -35.4 (39.0) | -28.1 (47.3)
Statistical Analysis 1: Comparison: TAS-303 3 mg vs Placebo; TAS-303 3 mg group vs. Placebo group for the mean percentage changes in IEF per 24 hours from baseline to Week 8; Test type: Superiority; p = 0.329, t-test, 2 sided; Mean Difference (Final Values) = -6.7, 95% CI 2-sided [-20.1 to 6.7], Standard Error of Mean 6.80
Statistical Analysis 2: Comparison: TAS-303 6 mg vs Placebo; TAS-303 6 mg group vs. Placebo group for the mean percentage changes in IEF per 24 hours from baseline to Week 8; Test type: Superiority; p = 0.285, t-test, 2 sided; Mean Difference (Final Values) = -7.3, 95% CI 2-sided [-20.9 to 6.2], Standard Error of Mean 6.84

3. Secondary Outcome: Incontinence Episode Frequency (IEF) Per 24 Hours at Baseline and Week 4
Time Frame: Baseline to Week 4 (4 weeks in treatment period)
Population: PPS was used for the analysis.
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | TAS-303 3 mg | TAS-303 6 mg | Placebo
Number analyzed (Participants) | 84 | 80 | 81
episodes
  IEF per 24 hours at baseline | 2.9 (2.3) | 2.5 (1.5) | 2.6 (1.7)
  IEF per 24 hours at Week 4: number analyzed (Participants) | 83 | 79 | 81
  IEF per 24 hours at Week 4 | 2.3 (2.2) | 2.0 (1.5) | 2.2 (1.7)

4. Secondary Outcome: Mean Percentage Changes in Incontinence Episode Frequency (IEF) Per 24 Hours From Baseline to Week 4
Time Frame: Baseline to Week 4 (4 weeks in treatment period)
Population: PPS was used for the analysis.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | TAS-303 3 mg | TAS-303 6 mg | Placebo
Number analyzed (Participants) | 83 | 79 | 81
Percentage change | -23.1 (37.3) | -23.9 (33.8) | -11.7 (45.4)
Statistical Analysis 1: Comparison: TAS-303 3 mg vs Placebo; TAS-303 3 mg group vs. Placebo group for the mean percentage changes in IEF per 24 hours from baseline to Week 4; Test type: Superiority; p = 0.082, t-test, 2 sided; Mean Difference (Final Values) = -11.3, 95% CI 2-sided [-24.1 to 1.5], Standard Error of Mean 6.48
Statistical Analysis 2: Comparison: TAS-303 6 mg vs Placebo; TAS-303 6 mg group vs. Placebo group for the mean percentage changes in IEF per 24 hours from baseline to Week 4; Test type: Superiority; p = 0.057, t-test, 2 sided; Mean Difference (Final Values) = -12.1, 95% CI 2-sided [-24.7 to 0.4], Standard Error of Mean 6.34

5. Secondary Outcome: Incontinence Episode Frequency (IEF) Per 24 Hours at Baseline and Week 4 in SUI Subgroup
Time Frame: Baseline to Week 4 (4 weeks in treatment period)
Population: PPS was used for the analysis. This analysis was conducted in SUI subgroup. This subgroup includes patients with only SUI but excludes those with MUI.
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | TAS-303 3 mg | TAS-303 6 mg | Placebo
Number analyzed (Participants) | 63 | 61 | 61
episodes
  IEF per 24 hours at baseline | 2.7 (2.4) | 2.5 (1.5) | 2.6 (1.7)
  IEF per 24 hours at Week 4: number analyzed (Participants) | 62 | 60 | 61
  IEF per 24 hours at Week 4 | 2.0 (1.9) | 1.9 (1.5) | 2.3 (1.9)

6. Secondary Outcome: Mean Percentage Changes in Incontinence Episode Frequency (IEF) Per 24 Hours From Baseline to Week 4 in SUI Subgroup
Time Frame: Baseline to Week 4 (4 weeks in treatment period)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | TAS-303 3 mg | TAS-303 6 mg | Placebo
Number analyzed (Participants) | 62 | 60 | 61
Percentage change | -26.5 (34.8) | -25.8 (33.5) | -8.9 (46.3)
Statistical Analysis 1: Comparison: TAS-303 3 mg vs Placebo; TAS-303 3 mg group vs. Placebo group for the mean percentage changes in IEF per 24 hours from baseline to Week 4; Test type: Superiority; p = 0.019, t-test, 2 sided; Mean Difference (Final Values) = -17.6, 95% CI 2-sided [-32.2 to -3.0], Standard Error of Mean 7.38
Statistical Analysis 2: Comparison: TAS-303 6 mg vs Placebo; TAS-303 6 mg group vs. Placebo group for the mean percentage changes in IEF per 24 hours from baseline to Week 4; Test type: Superiority; p = 0.023, t-test, 2 sided; Mean Difference (Final Values) = -16.9, 95% CI 2-sided [-31.5 to -2.3], Standard Error of Mean 7.36

7. Secondary Outcome: Incontinence Episode Frequency (IEF) Per 24 Hours at Baseline and Week 8 in SUI Subgroup
Time Frame: Baseline to Week 8 (8 weeks in treatment period)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | TAS-303 3 mg | TAS-303 6 mg | Placebo
Number analyzed (Participants) | 63 | 61 | 61
episodes
  IEF per 24 hours at baseline | 2.7 (2.4) | 2.5 (1.5) | 2.6 (1.7)
  IEF per 24 hours at Week 8 | 1.8 (2.1) | 1.8 (1.8) | 2.0 (2.0)

8. Secondary Outcome: Mean Percentage Changes in Incontinence Episode Frequency (IEF) Per 24 Hours From Baseline to Week 8 in SUI Subgroup
Time Frame: Baseline to Week 8 (8 weeks in treatment period)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | TAS-303 3 mg | TAS-303 6 mg | Placebo
Number analyzed (Participants) | 63 | 61 | 61
Percentage change | -37.4 (33.1) | -35.7 (37.8) | -26.1 (47.8)
Statistical Analysis 1: Comparison: TAS-303 3 mg vs Placebo; TAS-303 3 mg group vs. Placebo group for the mean percentage changes in IEF per 24 hours from baseline to Week 8; Test type: Superiority; p = 0.125, t-test, 2 sided; Mean Difference (Final Values) = -11.4, 95% CI 2-sided [-25.9 to 3.2], Standard Error of Mean 7.36
Statistical Analysis 2: Comparison: TAS-303 6 mg vs Placebo; TAS-303 6 mg group vs. Placebo group for the mean percentage changes in IEF per 24 hours from baseline to Week 8; Test type: Superiority; p = 0.221, t-test, 2 sided; Mean Difference (Final Values) = -9.6, 95% CI 2-sided [-25.1 to 5.9], Standard Error of Mean 7.80

9. Secondary Outcome: Percentages of the Patients With an Incontinence Amount of ≤ 2.0 g (Deemed Dryness) in the 1-hour Pad Test at Week 8 in the Treatment Period
Time Frame: At Week 8 in the treatment period
Population: PPS was used for the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | TAS-303 3 mg | TAS-303 6 mg | Placebo
Number analyzed (Participants) | 84 | 80 | 81
Participants | 25 | 27 | 13

10. Secondary Outcome: Patient Global Impression-Improvement (PGI-I) Rates at Baseline, Week 4 and Week 8
Description: PGI-I was used to evaluate the patients' impression of improvement of urinary incontinence.
  The improvement of PGI-I was defined as the selection of "Very much better", "Much better", or "A little better".
  The investigator or subinvestigator instructed patients to evaluate the improvement of urinary incontinence at the evaluation time point using the following 7-point scale: (1) "Very much better"; (2) "Much better"; (3) "A little better"; (4) "No change"; (5) "A little worse"; (6) "Much worse"; and (7) "Very much worse".
Time Frame: Baseline to Week 8 (8 weeks in treatment period)
Population: PPS was used for the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | TAS-303 3 mg | TAS-303 6 mg | Placebo
Number analyzed (Participants) | 84 | 80 | 81
Participants
  Baseline | 28 | 29 | 26
  Week 4 | 49 | 58 | 44
  Week 8 | 61 | 55 | 53

11. Secondary Outcome: Any Adverse Events
Description: For tabulation of adverse events, the terms of diagnosis recorded in the eCRFs were converted according to the Medical Dictionary for Regulatory Activities (MedDRA) ver. 20.1 and were expressed as preferred terms of MedDRA.
Time Frame: Baseline to Week 8 (8 weeks in treatment period)
Population: All treated population was used for the analysis. This analysis set includes all patients enrolled in the observation period who received at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | TAS-303 3 mg | TAS-303 6 mg | Placebo
Number analyzed (Participants) | 85 | 86 | 85
Participants
  Any adverse events | 31 | 20 | 26
  Palpitations | 1 | 0 | 0
  Vertigo | 0 | 0 | 1
  Sudden hearing loss | 0 | 0 | 1
  Abdominal pain lower | 1 | 0 | 0
  Constipation | 2 | 1 | 0
  Dental caries | 0 | 0 | 1
  Diarrhoea | 0 | 2 | 0
  Gastritis | 0 | 0 | 1
  Nausea | 0 | 1 | 0
  Stomatitis | 1 | 0 | 0
  Vomiting | 1 | 0 | 1
  Malaise | 0 | 1 | 0
  Pyrexia | 0 | 1 | 0
  Thirst | 1 | 1 | 0
  Allergy to arthropod bite | 0 | 1 | 0
  Bronchitis | 0 | 1 | 1
  Cystitis | 2 | 0 | 1
  Gingivitis | 0 | 0 | 1
  Herpes zoster | 1 | 0 | 1
  Hordeolum | 1 | 0 | 0
  Influenza | 1 | 0 | 0
  Nasopharyngitis | 9 | 4 | 8
  Otitis media | 1 | 0 | 0
  Periodontitis | 0 | 1 | 0
  Pyuria | 1 | 0 | 0
  Upper respiratory tract infection | 1 | 0 | 0
  Cystitis bacterial | 0 | 1 | 0
  Arthropod sting | 0 | 0 | 1
  Muscle injury | 1 | 0 | 0
  Radius fracture | 0 | 1 | 0
  Spinal compression fracture | 0 | 1 | 0
  Wound | 0 | 0 | 1
  Skin injury | 0 | 0 | 1
  Ear abrasion | 1 | 0 | 0
  Alanine aminotransferase increased | 2 | 0 | 0
  Aspartate aminotransferase increased | 1 | 0 | 0
  Blood creatine phosphokinase increased | 1 | 1 | 0
  Blood potassium increased | 0 | 1 | 0
  C-reactive protein increased | 1 | 1 | 1
  Electrocardiogram QT prolonged | 1 | 0 | 0
  Eosinophil count increased | 0 | 1 | 0
  White blood cell count increased | 1 | 0 | 0
  Liver function test increased | 1 | 0 | 0
  Dyslipidaemia | 1 | 0 | 0
  Decreased appetite | 0 | 2 | 0
  Arthralgia | 0 | 1 | 0
  Back pain | 1 | 0 | 1
  Musculoskeletal pain | 0 | 0 | 1
  Myalgia | 1 | 0 | 1
  Tenosynovitis | 0 | 0 | 1
  Headache | 0 | 2 | 0
  Sleep disorder | 1 | 0 | 0
  Proteinuria | 0 | 0 | 1
  Hypotonic urinary bladder | 0 | 0 | 1
  Cough | 0 | 2 | 0
  Upper respiratory tract inflammation | 1 | 0 | 0
  Oropharyngeal pain | 0 | 0 | 1
  Dermatitis atopic | 1 | 0 | 0
  Dermatitis contact | 0 | 0 | 1
  Eczema | 0 | 0 | 2
  Rash | 1 | 0 | 0
  Skin discomfort | 0 | 0 | 1
  Hypertension | 1 | 0 | 0

12. Secondary Outcome: Advese Events Occurring in ≥2% of Patients in Any Treatment Group During the Treatment Period
Description: as for outcome 11
Time Frame: Baseline to Week 8 (8 weeks in treatment period)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | TAS-303 3 mg | TAS-303 6 mg | Placebo
Number analyzed (Participants) | 85 | 86 | 85
Participants
  Nasopharyngitis | 9 | 4 | 8
  Cystitis | 2 | 0 | 1
  Constipation | 2 | 1 | 0
  Diarrhoea | 0 | 2 | 0
  Decreased appetite | 0 | 2 | 0
  Headache | 0 | 2 | 0
  Cough | 0 | 2 | 0
  Alanine aminotransferase increased | 2 | 0 | 0
  Eczema | 0 | 0 | 2

13. Secondary Outcome: Adverse Drug Reactions
Description: as for outcome 11
Time Frame: Baseline to Week 8 (8 weeks in treatment period)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | TAS-303 3 mg | TAS-303 6 mg | Placebo
Number analyzed (Participants) | 85 | 86 | 85
Participants
  Any Events | 6 | 0 | 0
  Constipation | 1 | 0 | 0
  Alanine aminotransferase increased | 1 | 0 | 0
  Aspartate aminotransferase increased | 1 | 0 | 0
  Blood creatine phosphokinase increased | 1 | 0 | 0
  White blood cell count increased | 1 | 0 | 0
  Liver function test increased | 1 | 0 | 0
  Rash | 1 | 0 | 0

14. Secondary Outcome: Serious Adverse Events
Time Frame: Baseline to Week 8 (8 weeks in treatment period)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | TAS-303 3 mg | TAS-303 6 mg | Placebo
Number analyzed (Participants) | 85 | 86 | 85
Participants | 0 | 0 | 0

15. Secondary Outcome: Adverse Events Leading to Discontinuation of Administration
Time Frame: Baseline to Week 8 (8 weeks in treatment period)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | TAS-303 3 mg | TAS-303 6 mg | Placebo
Number analyzed (Participants) | 85 | 86 | 85
Participants
  Any adverse events leading to discontinuation of administration | 0 | 1 | 0
  Radius fracture | 0 | 1 | 0
  Spinal compression fracture | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Baseline to Week 8 (8 weeks in treatment period)
Description: All treated population was used for the analysis. This analysis set includes all patients enrolled in the observation period who received at least 1 dose of the study drug.
Arm/Group | TAS-303 3 mg | TAS-303 6 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/86 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/86 | 0/85
Other Adverse Events (participants affected / at risk) | 31/85 | 20/86 | 26/85
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAS-303 3 mg (N=85) | TAS-303 6 mg (N=86) | Placebo (N=85)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Thirst (General disorders) | 1 (1) | 1 (1) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 9 (9) | 4 (4) | 8 (9)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cystitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ear abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotonic urinary bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin discomfort (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-08-16): https://cdn.clinicaltrials.gov/large-docs/83/NCT02906683/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/83/NCT02906683/SAP_001.pdf